CLINICAL TRIAL: NCT03713554
Title: Use of Functional Near-infrared Spectroscopy to Investigate Role of Human Auditory Cortex Plasticity and Multi-sensory Integration on Cochlear Implant Performance After Single-sided Deafness
Status: Withdrawn | Type: Observational
Why Stopped: Anticipated funding was never acquired to begin actual enrollment.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Gregory Basura, Otorhinolaryngology Department - Faculty and Staff Medical School - Faculty and Staff, University of Michigan
Other Study IDs: HUM00137093
Record Dates: First submitted 2018-10-10; First posted 2018-10-19 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Hearing Loss
Keywords: SSD, unilateral hearing loss
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Unilateral

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: FNIRS Observational — In addition to completing an Informed Consent and survey questions, fNIRS Imaging and Electroencephalography (EEG) will take place will take place:The fNIRS imaging is experimental technology that has not been approved by the FDA. EEG is a noninvasive way to record electrical activity of the brain. The recording device is made up of electrodes that are fixed to a snug-fitting elastic cap. An MRI and EEG will follow the fNIRS procedure. The MRI will be performed before participants undergo fNIRS or EEG. The MRI will be done to show there are no lesions in the inner ear and therefore is a recruitment clearance tool.

SUMMARY:
The timing of brain changes that may influence hearing rehabilitation within human A1 after single-sided deafness (SSD) is not known. The goal is to determine when A1 neural plasticity occurs following SSD onset.

DETAILED DESCRIPTION:
Sudden onset, profound unilateral sensorineural hearing loss, or single-sided deafness (SSD) is common (60,000 annually in US). Permanent SSD leads to listener disability and long-term challenges with sound localization and speech perception. The only definitive auditory rehabilitation for SSD is a cochlear implant (CI). Limited research on optimal timing for CI after SSD exists since insurance authorization typically requires bilateral deafness for CI placement. Secondly, limited CI compatible brain imaging technology exists to investigate changes pre- and post-CI in SSD. Thus, lack of systematic research results in random CI placement in SSD with inconsistent auditory performance that may be due, in part, to variable neural activation in primary auditory cortex (A1). Animal models and humans with SSD show enhanced A1 neural responses with sound stimulation of the remaining only-hearing ear1,2. Also, cross-modal plasticity3 (increased A1 neural responses to non-auditory sensory systems) leads to preferential A1 activation to somatosensory and visual stimuli4,5,6 in SSD. Essentially, non-auditory sensory systems "recruit" A1 neurons away to become responsive to new non-auditory stimulation. This limits the ability of A1 neurons to respond to auditory stimulation once CI rehabilitation is implemented. Importantly, a sensitive time window after SSD when these brain changes occur may impact A1 neural auditory responses and ultimately CI performance and speech perception.

Activation strength of A1 neurons is associated with optimal CI speech recognition and performance7,8. The investigators predict that if A1 neurons opposite SSD are kept active by increased sensitivity to only-hearing ear stimulation after SSD they would be less likely to be "reassigned" to non-auditory cross-modal plasticity. Alternatively, if only-hearing ear inputs to A1 are not sufficient, or if more somatosensory and/or visual inputs occur after SSD, fewer A1 neurons will be available to respond to CI stimulation and speech performance may suffer. The objective of these studies is first, to understand the timing and nature of both A1 cross-modal plasticity (sensitivity to somatosensory and/or visual systems) and only-hearing ear pathway enhancement in SSD. Second, is to examine the impact of CI on reversing these changes that may affect CI performance.

Human research on SSD and CI is sparse due to inadequate brain imaging technology that can measure A1 neural activity that is also CI compatible. Functional near-infrared spectroscopy (fNIRS) and event-related potentials (ERPs) with electroencephalography (EEG), when used together, can capture localization (fNIRS) and timing (EEG) of correlates of A1 neural responses (fNIRS) to distinguish between the effects of cross-modal and only-hearing ear stimulation pre- and post-CI. Using stimulation/silence block recording conditions in SSD adults, A1 hemodynamic responses (correlates of neural activity) and resting state functional cortical connectivity (RSFC; index of inter-cortical connections) will be measured with fNIRS and ERPs and correlated with only-hearing ear and cross-modal plasticity9,10 and CI speech performance11.

Specific Aim 1: Determine when A1 neural plasticity occurs following SSD onset. The timing of brain changes that may influence hearing rehabilitation within human A1 after SSD is not known. The goal of this aim is to identify plasticity that occurs when there is no CI intervention and characterize when A1 neurons are either influenced by only-hearing ear, somatosensory and/or visual inputs after SSD. Experiment 1. A1 hemodynamic responses (fNIRS correlate of neural activity) and changes in brain RSFC and ERPs to somatosensory, visual and only-hearing ear stimulation will be recorded 1, 3, 6, 9 and 12 months after SSD onset. The investigators predict cross-modal plasticity and A1 responses to only-hearing ear stimulation after SSD will have specific timing patterns of onset.

Specific Aim 2: Identify changes in A1 neural plasticity that follows CI rehabilitation.

The goal of this aim is to determine how and when CI placement affects A1 plasticity in SSD. As such, the investigators will determine when and if brain changes can be prevented that may hinder eventual CI performance. Experiment 2: Participants following CI placement that is either early- (<6mos), delayed- (6-12mos) or late- (>12mos-5yrs) after SSD and random insurance authorization will be analyzed for hemodynamic responses, changes in RSFC and ERPs to somatosensory, visual, CI, and only-hearing ear stimulation 1-12 months after CI. The investigators predict optimal CI speech performance will be associated with stronger fNIRS/ERP responses to early- and mid-CI placement that will reverse A1 responses to cross-modal stimulation.

Specific Aim 3: Identify neurocognitive profiles of successful CI rehabilitation of SSD. A1 plasticity pre- and post-CI and its relationship to speech performance in SSD will be measured. Experiment 3: CI speech performance testing will be conducted and results are expected to correlate with degrees/timing of plasticity from Aims 1 and 2. The investigators predict those with less A1 cross-modal plasticity and greater responses to the only-hearing ear will show better CI speech performance, while greater A1 responses to somatosensory and/or visual stimulation will perform more poorly with CI.

Clinical Significance: The investigators predict that this project will uncover timing and mechanisms of key auditory brain plasticity that follows adult-onset SSD and CI rehabilitation. This work will also demonstrate that fNIRS may prove to be a superior measure of A1 plasticity that could be used going forward to improve the timing of placement of CI for SSD to optimize speech performance and auditory rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 18

Exclusion Criteria:

* prior otologic surgery
* any SSD less than profound hearing loss
* any subjected treated at an outside institution

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SSD Patients
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hemodynamic activity (fNIRS correlate of neural activity) in primary auditory cortex (A1) other non-auditory (somatosensory and visual) after single sided deafness; before and after cochlear implantation (CI). | 12 months
  Functional near-infrared spectroscopy (fNIRS) is a non-invasive tool for measuring cortical hemodynamic activity in human auditory and non-auditory studies. fNIRS measures changing optical properties of the brain using infrared (IR) light to extrapolate and quantify hemodynamic responses through neurovascular coupling. When a specific brain region is activated, fNIRS measures changes in local hemoglobin as an index/correlate of neural activity within a chosen brain region.

SECONDARY OUTCOMES:
Resting state functional connectivity (RSFC; connectivity) between primary auditory cortex (A1) and other non-auditory (somatosensory and visual) cortices after single sided deafness; before and after cochlear implantation (CI). | All fNIRS recordings will be taken at baseline (Aim 1) 1,3,6,9 and 12 months after single-sided deafness and at the same intervals after CI (Aim 2).
  Resting state functional connectivity (RSFC) is the association of baseline activity between two brain regions. Although RSFC portends anatomical/structural interactions it does not assess activity at the individual neuron level. By assessing RSFC, we obtain information regarding spatiotemporal patterns of hemodynamic cortical responses across brain regions, which are thought to reflect plastic changes that play a role in both adaptive and maladaptive conditions. RSFC has been proposed to represent contextual influences of connections involved in local processing, connections between regions that are likely to work together in the future, or serve to coordinate neural activity.
Event-related potentials (ERPs from EEG recordings) in auditory cortex (A1) and other non-auditory (somatosensory and visual) cortices after single sided deafness; before and after cochlear implantation (CI) | All EEG recordings will be taken at baseline (Aim 1) 1,3,6,9 and 12 months after single-sided deafness and at the same intervals after CI (Aim 2).
  Electroencephalography (EEG) is another non-invasive method used to capture neuro-electric activity. Scalp electrodes measure currents that flow during excitation of cortical pyramidal neurons. EEG measures event-related potentials (ERPs) that are fluctuations time-locked to an event or stimulus onset. Many investigative approaches combine fNIRS for spatial resolution and EEG for temporal resolution as each is linked to the same neuronal activities and therefore complementary.
Cochlear implant (CI) speech performance | Cochlear implant speech performance will be measured 6 and 12 months after implantation (Aim 3).
  All CI participants will undergo formal speech recognition testing per the clinical standard of care. Measures commonly used in clinical care of participants with CIs will be used in this study. Consonant-Nucleus-Consonant (CNC) monosyllabic words will be presented at a level of 60dB sound pressure level (SPL) in quiet. Additionally, two lists of sentences from the Bamford-Kowal-Bench Speech-in-Noise-Test (BKB-SIN) will be administered according to recommendations of the Minimal Speech Test Battery and will determine the SNR at which participants understand 50% of the words in the sentences.

IPD SHARING:
Plan to Share IPD: Yes
The researcher is open to sharing data by an appropriate mechanism indicated by NIH program staff.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After scientific papers are accepted for publication, data will be available for 7 years after study completion.
Access Criteria: Researchers requesting data will first have to sign a data sharing agreement, agreeing to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, electronically securing the data while in use, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, no use of the data for commercial purposes and proper acknowledgement of the data resource.